CLINICAL TRIAL: NCT00793026
Title: Safety Dermatological Evaluation: Genital Mucous Irritation - Test in Use - Dermacyd Breeze Pocket BR (Lactic Acid).
Brief Title: Dermacyd Breeze Pocket BR (Lactic Acid) - Acceptability
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04365
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (1):
- 1 (Experimental): Dermacyd Breeze Pocket BR (Lactic Acid)
  Interventions: Drug: Dermacyd Breeze Pocket BR (Lactic Acid)

INTERVENTIONS:
Drug: Dermacyd Breeze Pocket BR (Lactic Acid) — Dermacyd Breeze Pocket BR (Lactic Acid) during 21 consecutive days

SUMMARY:
The purpose of this study is to prove the safety of the gynaecological formulation in normal conditions of use.

ELIGIBILITY:
Inclusion criteria:

* Integral skin test in the region;
* To use products of the same category;

Exclusion criteria:

* Lactation or gestation;
* Use of anti-inflammatory, anti-histaminic or immunosuppressant drugs;
* Cutaneous disease (local or spread) in the evaluation area;
* Pathology which may cause immunity depression, such as HIV, diabetes;
* Endocrine pathology
* Solar exposure 15 days before evaluation;
* Treatment until four months before the selection.
* Allergic or atopic history to cosmetics products

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Absence of irritation | Throughout the study
Good acceptability | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com